CLINICAL TRIAL: NCT07351071
Title: A Prospective, Multicenter, Single-arm, Post Market Study to Evaluate the Safety and Performance of the Signia™ Circular Stapler With Tri-Staple™ Technology in Elective Open or Minimally Invasive Left-sided Colon, Sigmoid, and Rectal Resections (SECURE)
Brief Title: Post-Market Study of the Signia Circular Stapler With Tri-Staple Technology in Left-sided Colon, Sigmoid, and Rectal Resections
Acronym: SECURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT24002
Record Dates: First submitted 2026-01-16; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Anastomosis; Left-sided Colon Resection; Anastomotic Leak; Anastomotic Complication; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Postoperative Complications; Anastomotic Leaks
Keywords: Colorectal Anastomosis; Left-sided Colon Resection; Circular stapler; Anastomotic Leak; Rectal cancer; Low anterior resection; Powered stapler
MeSH Terms: conditions — Anastomotic Leak; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases; Postoperative Complications; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Left sided colon/colorectal procedure with creation of an anastomosis (Experimental): single arm study, no control arm
  Interventions: Device: Signia™ circular stapler with Tri-Staple™ Technology (Signia™ Circular Stapling system)

INTERVENTIONS:
Device: Signia™ circular stapler with Tri-Staple™ Technology (Signia™ Circular Stapling system) — Signia™ Circular Stapling system used for the creation of an anastomosis

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the Signia™ power handle, Signia™ circular adapter, and Signia™ Tri-Staple™ 2.0 circular reloads (hereafter referred to as Signia™ circular stapler) in patients undergoing left sided colon, sigmoid, or rectal resections in a post market setting.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and performance of the Signia™ circular stapler, for the creation of anastomoses assessed by the incidence of anastomotic leak within 30 days following use in subjects undergoing left sided colon, sigmoid, or rectal resections.

The secondary objectives of this study are to assess safety and performance outcomes within 90 days following the use of the Signia™ circular stapler in subjects undergoing left sided colon, sigmoid, or rectal resections.

ELIGIBILITY:
Preoperative Inclusion Criteria:

1. Subject is competent and willing to provide documented informed consent to participate in this clinical study
2. Subject is intended to undergo an elective left sided colon/colorectal procedure where a creation of an anastomosis will be completed with the Signia™ circular stapler
3. Subject is ≥ 18 years of age at time of consent

Preoperative Exclusion Criteria:

1. Subject is unable or unwilling to comply with the study requirements or follow-up schedule
2. Subject with ASA classification ≥ IV
3. Subject is pregnant (as determined by standard site practices)
4. The procedure is an emergency procedure
5. The procedure is a revision/reoperation for the same indication
6. The subject has a documented confounding medical condition which in the opinion of the investigator, will not be appropriate for the study, or the subject has an estimated life expectancy of less than 6 months
7. Subject has participated or plans to participate in an investigational drug or device research study that would interfere with the results of this study
8. Subject will undergo multiple synchronous colon resections
9. Subject with a bleeding disorder or is undergoing anticoagulant treatment that has not been reversed (anticoagulant prophylaxis prescribed as part of the surgical protocol is allowed)
10. Subject has undergone chemotherapy or received biologics within 6 weeks prior to the day of the procedure
11. Subject has history of chronic corticosteroid use (used greater than 3 months within a year prior to the index procedure)
12. Subject has chronic immunosuppression therapy (used greater than 3 months within a year prior to the index procedure)
13. Any subject undergoing an ileal-anal pouch anastomosis surgery

Intraoperative Exclusion Criteria

1. Anastomosis not attempted with the Signia™ circular stapler
2. Any subject for which the device is intended to be used outside the instructions for use (IFU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of anastomotic leak | within 30 days, +/- 14 days
  Incidence of anastomotic leak following the use of the Signia™ circular stapler used in subjects undergoing left sided colon, sigmoid, or rectal resections. Diagnosis will be confirmed postoperatively by computed tomography (CT) imaging (with or without a contrast agent), or postoperatively via direct verification during re-operation. Anastomotic leakage confirmed to have occurred at a staple line other than the colon/colorectal anastomosis created with the Signia™ circular stapler will not impact the primary endpoint analysis.

SECONDARY OUTCOMES:
Incidence of anastomotic leaks | within 90 days, +/- 14 days
  Incidence of anastomotic leak following the use of the Signia™ circular stapler used in subjects undergoing left sided colon, sigmoid, or rectal resections. Diagnosis will be confirmed postoperatively by computed tomography (CT) imaging (with or without a contrast agent), or postoperatively via direct verification during re-operation. Anastomotic leakage confirmed to have occurred at a staple line other than the colon/colorectal anastomosis created with the Signia™ circular stapler will not impact the primary endpoint analysis.
Clinical significance of anastomotic leaks | within 90 days, +/- 14 days
  Anastomotic leaks graded according to International Study Group of Rectal Cancer (ISGRC):
  Grade A: Anastomotic leakage results in no change in patients' management. Grade B: Leakage requires active therapeutic intervention but is manageable without re-laparotomy/operative intervention*.
  Grade C: Anastomotic leakage requires re-laparotomy/operative intervention*.
  *Operative intervention was added to the ISGRC definition for the purpose of this study.
Incidence of a Signia™ circular stapler and accessory components device deficiency (DD) | Day 0 (day of surgery)
  Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance.
Incidence of anastomotic bleeding | within 30 and 90 days, +/- 14 days
  bleeding at the anastomotic site that requires endoscopic or surgical intervention
Incidence of device-related adverse events | within 90 days, +/- 14 days
  Adverse events related to Signia™ circular stapler and accessory components. An adverse event is defined as "Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device and whether anticipated or unanticipated."
Length of hospital stay | discharge (post-surgery up to 90 days, +/- 14 days)
  Length of hospital stay for the index procedure (from admission to discharge) after the Signia™ circular stapler was used in subjects undergoing left sided colon, sigmoid, or rectal resections
Incidence of re-operation or surgical intervention | within 90 days, +/- 14 days
  Incidence of re-operation or surgical intervention due to an adverse event related to the Signia™ circular stapler or accessory components

OTHER OUTCOMES:
Surgeon satisfaction | Day 0 (day of surgery)
  Surgeon satisfaction via a questionnaire
Incidence of serious device-related adverse events | within 90 days, +/- 14 days
  serious device-related adverse events related to Signia™ circular stapler and accessory components. A serious adverse event is defined as an "Adverse event that led to any of the following:
  1. Death,
  2. Serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function including chronic diseases, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function, or
  3. foetal distress, foetal death, a congenital abnormality, or birth defect including physical or mental impairment.
Clavien-Dindo classification of surgical complications | within 90 days, +/- 14 days
  Clavien-Dindo classification of postoperative device related adverse events and serious device related adverse events.
Readmission to hospital | within 30 and 90 day, +/- 14 days
  Readmission to hospital for study index procedure-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Louise Jackson, MD, FACS, MBBS, MA, Principal Investigator — Duke Raleigh Hospital; John Monson, MD, FACS, Principal Investigator — Northwell Health
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No